CLINICAL TRIAL: NCT00657657
Title: Immune Response to a Hepatitis B Vaccine Challenge Dose in Healthy Subjects Who Received Primary Vaccination of GlaxoSmithKline Biologicals' Hepatitis B Vaccine, Approximately 20 Years Ago.
Brief Title: Safety and Immunogenicity of a Booster Dose of GlaxoSmithKline (GSK) Biologicals' Hepatitis B Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 110071
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Results first posted 2009-09-14 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-10

CONDITIONS: Hepatitis B
Keywords: Hepatitis; vaccine
MeSH Terms: conditions — Hepatitis B; Hepatitis

ARMS (4):
- Group 1 (Experimental): Neonates from mother HBsAg (+) and HBeAg (+) had received HBV vaccine at Month 0, 1, 2, 12, 60 (5 doses)
  Interventions: Biological: Engerix™-B
- Group 2 (Experimental): Neonates from mother HBsAg (+) and HBeAg (+) had received HBV vaccine at Month 0, 1, 2, 12 (4 doses)
  Interventions: Biological: Engerix™-B
- Group 4 (Experimental): Neonates from mother HBsAg (+) and HBeAg (-) had received HBV vaccine at Month 0, 1, 2, 12 (4 doses)
  Interventions: Biological: Engerix™-B
- Group 6 (Experimental): Neonates from mother HBsAg (-) and HBeAg (-) had received HBV vaccine at Month 0, 1, 2, 12 (4 doses)
  Interventions: Biological: Engerix™-B

INTERVENTIONS:
Biological: Engerix™-B — A challenge dose of hepatitis B vaccine will be administered to all subjects as a deep intramuscular injection in the deltoid region of the non-dominant arm.

SUMMARY:
In this study, subjects who received primary neonatal vaccination with hepatitis B vaccine at 0, 1, 2, 12 months, 20 years ago in the 103860/272 primary study will be evaluated for immunological memory to hepatitis B vaccine via assessment of the response to a vaccine challenge dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female adult who received the complete neonatal primary vaccination course of hepatitis B vaccine (Engerix™-B), in the 103860/272 primary study approximately 20 years earlier.
* Documented level of anti-HBs antibody concentrations < 100 milli-international units per milliliter (mIU/ml) at the previous long-term time-point for which serological results are available for that subject.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the hepatitis B challenge dose.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the hepatitis B vaccine challenge dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before the hepatitis B vaccine challenge dose and ending 30 days after.
* Subjects who received a booster dose of hepatitis B vaccine outside the context of this study between the long-term time-point at the documented level of anti-HBs antibody concentrations and the current challenge dose study visit.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* Acute disease at the time of enrolment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Administration of immunoglobulins and/or any blood products within the three months preceding the hepatitis B vaccine challenge dose or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Poovorawan Y et al. Persistence of anti-HBs antibodies and immune memory 20-years after hepatitis B vaccination among children in Thailand. Abstract presented at the 9th International Congress of Tropical Pediatrics (ICTP). Bangkok, Thailand. 18-20 October 2011.
- [Derived] Poovorawan Y, Chongsrisawat V, Theamboonlers A, Crasta PD, Messier M, Hardt K. Long-term anti-HBs antibody persistence following infant vaccination against hepatitis B and evaluation of anamnestic response: a 20-year follow-up study in Thailand. Hum Vaccin Immunother. 2013 Aug;9(8):1679-84. doi: 10.4161/hv.24844. Epub 2013 May 31. PMID 23732904
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 110071 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110071 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110071 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110071 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110071 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110071 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who received primary neonatal Engerix™-B vaccination 20 years ago in the 103860/272 primary study and who had anti-hepatitis B surface antigen (HBs) antibody concentrations < 100 milli-international units per milliliter (mIU/ml) at the previous available long-term time-point (NCT00240539), were invited to participate in the current study.
Groups:
- Engerix Group: Subjects received a challenge dose of hepatitis B vaccine (Engerix™-B).
Period: Overall Study
Arm/Group | Engerix Group
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Engerix Group
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.9 (0.35)
Gender [Count of Participants; unit: Participants]
  Female | 19
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With an Immune Response to a Challenge Dose of Hepatitis B Vaccine
Description: Immune response to a challenge dose of hepatitis B vaccine is defined as
  * at least a 4-fold rise in post-challenge dose anti-HBs antibody concentrations in subjects seropositive (≥ 3.3 mIU/mL) at the previous available long-term time point, or
  * a post-challenge dose anti-HBs antibody concentrations ≥ 10 mIU/mL in subjects seronegative (<3.3 mIU/mL) at the previous available long-term time point.
Time Frame: One month after the hepatitis B vaccine challenge dose
Measure: Number; unit: subjects
Arm/Group | Engerix Group
Number analyzed (Participants) | 29
subjects | 28

2. Secondary Outcome: Number of Subjects With Anti-HBs Antibody Concentrations Above Pre-defined Cut-off Values
Description: Anti-hepatitis B surface antigen (anti-HBs) antibody cut-off values assessed include 3.3, 10 and 100 mIU/mL.
Time Frame: One month after the hepatitis B vaccine challenge dose
Measure: Number; unit: subjects
Arm/Group | Engerix Group
Number analyzed (Participants) | 29
subjects
  ≥3.3 mIU/mL | 29
  ≥10 mIU/mL | 28
  ≥100 mIU/mL | 27

3. Secondary Outcome: Concentration of Anti-HBs Antibodies
Description: Concentrations are given as Geometric Mean Concentrations (GMCs), calculated on subjects seropositive (subjects with anti-HBs antibody concentrations ≥ 3.3 mIU/mL) post-challenge dose.
Time Frame: One month after the hepatitis B vaccine challenge dose
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Engerix Group
Number analyzed (Participants) | 29
mIU/mL | 1082.4 [561.0 to 2088.6]

4. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events
Description: An adverse event is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: During the 31-day follow-up period after the challenge dose of hepatitis B vaccine
Measure: Number; unit: subjects
Arm/Group | Engerix Group
Number analyzed (Participants) | 29
subjects | 0

5. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events
Description: A serious adverse event is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: During the 31-day follow-up period after the challenge dose of hepatitis B vaccine
Measure: Number; unit: subjects
Arm/Group | Engerix Group
Number analyzed (Participants) | 29
subjects | 0

ADVERSE EVENTS:
Arm/Group | Engerix Group
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.